CLINICAL TRIAL: NCT07065903
Title: Nimodipine Systemic Exposure and Outcomes Following Aneurysmal Subarachnoid Hemorrhage: A Prospective Multi-centre Observational Study (ASH-II Study)
Brief Title: Nimodipine Variability in SAH
Acronym: ASH-II
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Health services (Other); Foothills Medical Centre (Other); Montreal Neurological Institute and Hospital (Other); University Health Network, Toronto (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Sherif Mahmoud, Associate Professor, University of Alberta
Other Study IDs: Pro00085618
Record Dates: First submitted 2025-07-02; First posted 2025-07-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Subarachnoid Aneurysm Hemorrhage; Subarachnoid Hemorrhage, Aneurysmal
Keywords: nimodipine; subarachnoid hemorrhage; pharmacokinetics
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aneurysmal subarachnoid hemorrhage (SAH) Patients: Adult patients admitted for aneurysmal SAH to any of the participating centres, who consent to participate in the study and meet the inclusion and exclusion criteria.

SUMMARY:
Aneurysmal subarachnoid hemorrhage (SAH) is a life-threatening neurological illness: it is bleeding in the brain after a bulging blood vessel (a brain aneurysm) ruptures. Although SAH accounts for only 5% of all strokes, it often happens in middle age and it puts a significant burden on many patients during their most productive years. Complications following SAH are common, and they can cause major long-term disability. Only one medication - nimodipine - has been proven to benefit the health and wellbeing of these patients. All SAH patients should receive nimodipine for 21 days at a fixed dose. However, our early work suggested that all patients are not getting equal amounts of nimodipine into their blood. In addition, the two different forms (structural mirror images) of nimodipine might have different effects. Reduced amounts of nimodipine in the blood may lessen its benefit and contribute to worsening health and wellbeing of SAH patients.

The overall goal of this research is to see what happens with different nimodipine doses and to confirm whether the two forms of nimodipine have different effects. The investigators will conduct a multi-centre study in adult patients admitted for SAH in Canada and the USA. The investigators will collect blood samples to determine the amount of each type of nimodipine in each participant's body, and then will check to see how each participant is doing at 90 days following SAH. They will also check other factors affecting nimodipine levels, so that they can in the future suggest dose recommendations that are actually tailored to each patient.

DETAILED DESCRIPTION:
Background and Importance:

Aneurysmal subarachnoid hemorrhage (SAH) is a life-threatening neurological illness characterized by the extravasation of blood into the subarachnoid space secondary to a ruptured brain aneurysm. Although SAH accounts for only 5% of all strokes, it often places a significant burden on the most productive years of a patient's life because of the relatively young average age at onset. Cerebral vasospasm and delayed cerebral ischemia (DCI) are common complications following SAH and are significant contributors to disability in those surviving the initial bleed. Several agents have been tested to target vasospasm and DCI, but nimodipine was the only drug therapy that was shown to significantly improve neurological outcomes, and current guidelines recommend that all patients receive fixed-dose racemic nimodipine for 21 days following ictus. However, the pilot data suggested significant variability of nimodipine concentrations in the plasma, but it was not clear if minimal or lack of systemic exposure to nimodipine denies its benefit and contributes to worsening patient outcomes. Furthermore, the investigators' pilot data suggested that the two enantiomers of nimodipine might have differential effects, but it was not clear if one enantiomer is preferred over the other.

The overall goal of this research is to characterize the predictors and the clinical consequences of altered exposure to nimodipine enantiomers in SAH patients.

Research Aims:

1. To determine the associations between systemic exposure to the two nimodipine enantiomers and the primary and secondary outcomes in SAH patients.
2. To determine whether nimodipine enantiomers differ in their effects on safety in SAH patients.
3. To determine the population pharmacokinetics of nimodipine enantiomers and to develop individualized dosing recommendations in SAH populations.

Approach:

This study is for a multi-centre prospective study in adult patients admitted to the hospital for SAH. Participants will have blood samples collected for the determination of plasma concentrations of nimodipine enantiomers. Participant data will be collected prospectively, and the primary outcome will be their modified Rankin Scale (mRS) score at 90 days following SAH onset. The mRS is a functional outcome scale commonly used SAH studies. Regression modeling will be used to determine if systemic exposures to nimodipine enantiomers (quantified as the area under the concentration-time curves) are independent predictors of mRS outcomes. Predictors of exposure to nimodipine enantiomers will also be determined using population pharmacokinetics, and individualized dosage regimens will be recommended.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years
* Diagnosis of aneurysmal SAH
* Provision of informed consent
* Treated with nimodipine
* Presence of intravascular catheter at the time of sampling

Exclusion Criteria:

* Anticipated hospital length of stay <48 hours
* Non-aneurysmal SAH
* Not treated with nimodipine
* Incarceration
* Delayed presentation to the hospital (>96 h from SAH onset)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted for SAH to any of the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score | 90 days from hospital admission
  The mRS is a measure of disability ranging from 0 (no symptoms) to 6 (death) and is the recommended functional outcome scale in studies involving SAH patients.

SECONDARY OUTCOMES:
Delayed Cerebral Ischemia (DCI) | 21 days from hospital admission
  DCI is defined as "the occurrence of focal neurological impairment or a decrease of at least 2 points on the GCS. Such changes are not apparent immediately after aneurysm occlusion and cannot be attributed to other causes"
Vasospasm | 21 days from hospital admission
  Vasospasm is defined as the presence of angiographic evidence of cerebral arterial narrowing

CONTACTS AND LOCATIONS:
Locations (3):
- VCU Medical Center, Richmond, Virginia, United States
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - University Health Network - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared in accordance with maintaining patient confidentiality.

REFERENCES:
- [Background] Lethaby A, Irvine G, Cameron I. Cyclical progestogens for heavy menstrual bleeding. Cochrane Database Syst Rev. 2000;(2):CD001016. doi: 10.1002/14651858.CD001016. PMID 10796587
- [Background] Vergouwen MD, Vermeulen M, van Gijn J, Rinkel GJ, Wijdicks EF, Muizelaar JP, Mendelow AD, Juvela S, Yonas H, Terbrugge KG, Macdonald RL, Diringer MN, Broderick JP, Dreier JP, Roos YB. Definition of delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage as an outcome event in clinical trials and observational studies: proposal of a multidisciplinary research group. Stroke. 2010 Oct;41(10):2391-5. doi: 10.1161/STROKEAHA.110.589275. Epub 2010 Aug 26. PMID 20798370
- [Background] Mahmoud SH, Ji X, Isse FA. Nimodipine Pharmacokinetic Variability in Various Patient Populations. Drugs R D. 2020 Dec;20(4):307-318. doi: 10.1007/s40268-020-00322-3. PMID 32902829
- See also: Neuro-CPK Laboratory Website — https://www.neuro-cpk-lab.com/